CLINICAL TRIAL: NCT01131585
Title: A 12-month, Two-armed, Randomized, Double-masked, Multicenter, Phase IIIb Study Assessing the Efficacy and Safety of Laser Photocoagulation as Adjunctive to Ranibizumab Intravitreal Injections vs. Laser Photocoagulation Monotherapy in Patients With Visual Impairment Due to Diabetic Macular Edema Followed by a 12 Month Follow up Period
Brief Title: Safety and Efficacy of Ranibizumab in Diabetic Macular Edema
Acronym: RELATION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: European drug approval.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002DDE13; 2010-018852-29 (EudraCT Number)
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Visual Impairment Due to Diabetic Macular Edema
Keywords: Diabetic macular edema; DME; Proliferative diabetic retinopathy; PDR; ranibizumab; laser
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Active laser photocoagulation and ranibizumab (Experimental): Active laser treatment applied at baseline and reapplied if needed at intervals no shorter than 3 months from the last treatment.
  Ranibizumab intravitreal injection given at baseline, at 30, 60 and 90 days and if needed, reapplied at intervals no shorter than 28 days from last treatment.
  Interventions: Procedure: Active laser photocoagulation; Drug: Ranibizumab 0.5 mg
- Active laser photocoagulation and sham injection (Active Comparator): Active laser treatment applied at baseline and reapplied if needed at intervals no shorter than 3 months from the last treatment.
  Sham intravitreal injection given at baseline, at 30, 60 and 90 days and if needed, reapplied at intervals no shorter than 28 days from last treatment.
  Interventions: Procedure: Active laser photocoagulation; Drug: Sham injections

INTERVENTIONS:
Procedure: Active laser photocoagulation — Active laser photocoagulation procedure at baseline and reapplied if needed at intervals no shorter than 3 months from the last treatment.
Drug: Sham injections — Sham intravitreal injections at baseline, 30, 60 and 90 days and if needed, reapplied at intervals no shorter than 28 days from last treatment.
  Arms: Active laser photocoagulation and sham injection
Drug: Ranibizumab 0.5 mg — Ranibizumab 0.5 mg/0.05 ml intravitreal injection at baseline, 30, 60 and 90 days and if needed, reapplied at intervals no shorter than 28 days from last treatment.
  Arms: Active laser photocoagulation and ranibizumab

SUMMARY:
This study was designed to confirm the efficacy and safety of laser photocoagulation as adjunctive therapy to ranibizumab 0.5 mg versus laser monotherapy in patients with visual impairment due to Diabetic Macular Edema. A subgroup of patients with Proliferative Diabetic Retinopathy were included to evaluate the efficacy and safety of laser photocoagulation as adjunctive therapy to ranibizumab 0.5 mg versus laser monotherapy in this population.

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity impairment caused by macular edema in at least one eye
* Type 1 or type 2 diabetes mellitus
* Stable medication of diabetes in past 3 month

Exclusion Criteria:

* Patients with uncontrolled systemic or ocular diseases
* Laser photocoagulation in the study eye for the last 3 months
* Any history of any intraocular surgery in the study eye within the past 3 months
* Blood pressure > 160/100 mmHg

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (34):
- Germany (34):
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Eichstätt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Landshut
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Mühlheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Postdam
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rosenheim
  - Novartis Investigative Site, Siegburg
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg

REFERENCES:
- See also: Click here for more information about this study: — http://www.NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants did not complete study due to early termination. Study was terminated because of drug approval.
Groups:
- Active Laser Photocoagulation and Ranibizumab: Active laser treatment applied at baseline and reapplied if needed at intervals no shorter than 3 months from the last treatment.
  Ranibizumab intravitreal injection given at baseline, 30, 60 and 90 days and if needed, reapplied at intervals no shorter than 28 days from last treatment.
- Active Laser Photocoagulation and Sham Injection: Active laser treatment applied at baseline and reapplied if needed at intervals no shorter than 3 months from the last treatment.
  Sham intravitreal injection given at baseline, 30, 60 and 90 days and if needed, reapplied at intervals no shorter than 28 days from last treatment.
Period: Overall Study
Arm/Group | Active Laser Photocoagulation and Ranibizumab | Active Laser Photocoagulation and Sham Injection
Started | 85 | 43
Completed | 0 | 0
Not Completed | 85 | 43
Not completed — Adverse Event | 0 | 2
Not completed — Abnormal laboratory value | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative problems | 1 | 1
Not completed — Study termination | 78 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Laser Photocoagulation and Ranibizumab | Active Laser Photocoagulation and Sham Injection | Total
Number analyzed (Participants) | 85 | 43 | 128
Age Continuous [Mean (Standard Deviation); unit: years]
  >=18 years | 63.5 (9.3) | 63.5 (10.5) | 63.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 16 | 48
  Male | 53 | 27 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change in Best-Corrected Visual Acuity (BCVA) From Baseline to Month 12
Description: Mean change in Best-Corrected Visual Acuity (BCVA) letters at 12 months compared to baseline was measured using Visual acuity (VA). VA accounts for the number of letters a participant can see using Early Treatment Diabetic Retinopathy Study (EDTRS)-like visual acuity testing charts, from a sitting position at a testing distance of 4 meters. BCVA means that the participant's refraction is already taken into account when VA is determined. A higher BCVA number at 12 months in reference to baseline indicates improved BCVA.
Time Frame: 12 months
Population: Full Analysis Set consisted of all participants who received at least one application of study treatment and had at least one post-baseline assessment for BCVA. No patient completed the 12 months observational period due to study early termination; therefore, the last observation carried forward (LOCF) method was used with data from 11.1 months.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Active Laser Photocoagulation and Ranibizumab | Active Laser Photocoagulation and Sham Injection
Number analyzed (Participants) | 85 | 43
Letters | 6.5 (8.6) | 1.4 (7.3)

ADVERSE EVENTS:
Arm/Group | Active Laser Photocoagulation and Ranibizumab | Active Laser Photocoagulation and Sham Injection
Serious Adverse Events (participants affected / at risk) | 14/85 | 5/43
Other Adverse Events (participants affected / at risk) | 32/85 | 10/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Laser Photocoagulation and Ranibizumab (N=85) | Active Laser Photocoagulation and Sham Injection (N=43)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 1
DIABETIC RETINAL OEDEMA (Study eye) (Eye disorders) | 1 | 0
DIABETIC RETINOPATHY (Fellow eye) (Eye disorders) | 1 | 0
RETINAL DETACHMENT (Fellow eye) (Eye disorders) | 0 | 2
VITREOUS HAEMORRHAGE (Fellow eye) (Eye disorders) | 0 | 1
ANAL SPHINCTER ATONY (Gastrointestinal disorders) | 1 | 0
CONCOMITANT DISEASE PROGRESSION (General disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
DIABETIC FOOT (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 0
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
THROMBOPHLEBITIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Laser Photocoagulation and Ranibizumab (N=85) | Active Laser Photocoagulation and Sham Injection (N=43)
EYE IRRITATION (Study eye) (Eye disorders) | 5 (5) | 0 (0)
EYE PAIN (Study eye) (Eye disorders) | 13 (13) | 4 (4)
LACRIMATION INCREASED (Study eye) (Eye disorders) | 5 (5) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 13 (13) | 6 (6)
HEADACHE (Nervous system disorders) | 5 (5) | 1 (1)
HYPERTENSION (Vascular disorders) | 4 (4) | 4 (4)

LIMITATIONS AND CAVEATS:
Early study termination due to European drug approval.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.